CLINICAL TRIAL: NCT03958357
Title: Multi-center Prospective Observational Clinical Follow-Up Study Advanced Gynecological Applicator - Venezia Configuration
Brief Title: Post Market Clinical Follow-up Study Venezia
Status: Completed | Type: Observational
Sponsor: Nucletron Operations BV (Industry)
Collaborators: Factory CRO (Industry)
Responsible Party: Sponsor
Other Study IDs: Venezia-CIP-001
Record Dates: First submitted 2019-05-06; First posted 2019-05-22 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2020-09

CONDITIONS: Cervical Cancer
Keywords: Cervix; Uterus; Vagina; Cancer; Gynecology; Cervical cancer; External beam radiation therapy; Brachytherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment arm: Single arm study, 40 participants will undergo brachytherapy with the Advanced Gynecological Applicator Venezia Configuration
  Interventions: Device: Advanced Gynecological Applicator configuration

INTERVENTIONS:
Device: Advanced Gynecological Applicator configuration — The Advanced Gynecological Applicator Venezia configuration is a gynaecological applicator for intracavitary and interstitial brachytherapy. The applicator consists of tubes, caps and templates to place needles, which can be combined to reach a wide range of target areas. The tubes and possibly used needles, guide the radioactive source of the afterloader to the target volume. Dose optimization and dose fractionation is performed with the goal of adapting the dose to the target volume without exceeding the dose volume constraints for the surrounding normal tissues according to the standard cervical cancer treatment of the centre.

SUMMARY:
The investigational device is the Advanced Gynecological Applicator (AGA) Venezia configuration, an applicator to treat locally advanced stage cervical cancer. The goal of the study is to assess the performance and the unknown risks or complications of the AGA Venezia configuration during clinical use of the applicator.

DETAILED DESCRIPTION:
This is a multi-center, prospective, post-market clinical follow-up study to assess the performance and the unknown risks or complications of the Advanced Gynecological Applicator (AGA) Venezia configuration during clinical use of the applicator. The AGA Venezia configuration is a CE-marked, FDA approved and commercially available product. The AGA Venezia configuration is a gynaecological applicator for intracavitary and interstitial brachytherapy. The radiation oncologist can use it for treatment of cancers in the vagina, cervix and uterus. Forty (40) participants will be included in this study at 5 sites: 3 centers in Europe and 2 centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced cervical cancer stage IB to IVA
* Patients eligible for brachytherapy according to the criteria of the treating radiation oncologist and center guidelines
* Patients that are eligible to undergo brachytherapy with the Advanced Gynecological Applicator Venezia Configuration according to the criteria of the treating radiation oncologist
* Patient is able to understand and has voluntarily signed and dated the Ethics Committee approved informed consent form prior to initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Patients that have been treated or will be treated for cancer other than cervical cancer.
* Advanced stage cervical cancer patients who have been treated with pelvic radiotherapy, incl. brachytherapy, before.
* Patients younger than 18 years at the time of diagnosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants with cervical cancer
Study Population: Participants will be included in this study at 5 centers: 3 centers in Europe and 2 centers in the United States. For all participants chemoradiation treatment is planned with curative intent. Since chemoradiation including external beam radiation therapy and brachytherapy is standard of care for these patients, patients are selected according to the clinical practice guidelines of the clinical center. The treating radiation oncologist decides which patients will undergo the brachytherapy with the Advanced Gynecological Applicator Venezia Configuration.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Performance of the AGA Venezia configuration applicator as assessed by the 'Applicator Performance Questionnaire' | Within one week after each individual insertion. No change is assessed. The procedure is performed per hospital standard. On average, the procedure and applicator insertions are performed twice.
  Performance of the device is assessed via the 'Applicator Performance Questionnaire' completed by the radiation oncologist. Scale is as follows: Completely Agree/Agree/Neutral/Disagree/Completely Disagree/Not Applicable. The primary endpoint, the third question ('I am able to deliver conformal dose to the tumor target volume while effectively avoiding the organs at risk') on the Questionnaire will be summarized through descriptive statistics in general summary tables. Additionally, responses will be recoded numerically ('Completely agree' = 1, 'Agree' = 2, 'Neutral' = 3, 'Disagree' = 4, and 'Completely disagree' = 5). A five-number summary (min, first quartile, median, third quartile and max) and a boxplot will be shown. The question will also be recoded as success ('Completely agree'&'Agree') and failure ('Neutral', 'Disagree' & 'Completely disagree').

SECONDARY OUTCOMES:
Risks and/or complications of the AGA Venezia configuration applicator as assessed by the 'Risks and Complications Questionnaire' | Immediately after each insertion and followed up during the first follow-up visit, typically three months after the last insertion. The procedure is performed per hospital standard. On average, the procedure and applicator insertions are performed twice.
  Unknown risks or complications are assessed via the 'Risks and Complications Questionnaire' completed by the treating radiation oncologist. The treating radiation oncologist will be asked to complete this questionnaires to assess whether risks and complications occurred or not. There is no scale, but answer options include yes/no. The value "NO" is considered a better outcome. "YES" constitutes the worst outcome. Descriptive statistics presented in general summary tables will be provided, summarizing the number of non-missing observations (n), mean, standard deviation, minimum, median and maximum for quantitative data. For categorical data, frequency counts and percentages will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Ina Jurgenliemk-Schulz, MD, PhD, Principal Investigator — UMC Utrecht; Alina Sturdza, MD, Principal Investigator — Medical University Vienna; Robert Hobbs, MD, Principal Investigator — Johns Hopkins University; Elizabeth Harris, MD, Principal Investigator — University Hospital Case Western; Stefanie Corradini, Dr. med., Principal Investigator — Ludwig-Maximilians - University of Munich; Ina Jurgenliemk-Schulz, MD, PhD, Study Chair — UMC Utrecht; Christian Kirisits, Prof. Dr., Study Chair — Medical University Vienna
Locations (3):
- Medical University Vienna, Vienna, Austria
- Ludwig-Maximilians - University of Munich, Munich, Germany
- University Medical Centre Utrecht, Utrecht, Netherlands